CLINICAL TRIAL: NCT06906471
Title: A Single-Arm, Blinded, Fluorescent PSMA Histopathology Trial of AS1986NS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antelope Surgical Solutions, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 173786_007_1
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Cancer (Adenocarcinoma); Fluorescence Imaging
Keywords: fluorescent agent; PSMA; prostate surface membrane antigen; histopathology; fluorescence-guided surgery
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose of AS1986NS (Experimental): Single dose of AS1986NS administered as an injection through peripheral intravenous access.
  Interventions: Drug: AS1986NS

INTERVENTIONS:
Drug: AS1986NS — Single dose, IV, 100 µg of AS1986NS

SUMMARY:
A Single-Arm, blinded, fluorescent PSMA histopathology trial of AS1986NS

ELIGIBILITY:
Inclusion Criteria:

* suspected prostate cancer warranting standard of care multi-core prostate biopsy

Exclusion Criteria:

* Patients receiving same-day therapeutic Lutetium-177 or Actinium-225 PSMA receptor radiation isotope therapy treatment
* Patients with pre-existing, impaired or abnormal hepatic function, renal function, cardiac function, and abnormal elevated temperature
* Patients with a creatinine clearance cutoﬀ (CrCl) of < 60 mL/min

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of AS1986NS | Enrollment to 30 days post single infusion
  Demonstrate that AS1986NS is 'safe' as a microdosed <100 µg, <100 µL, 1 mg/mL per patient dose when introduced intravenously as a bolus through peripheral intravenous access by evaluation of the Adverse Events (AEs), including Serious Adverse Events (SAEs), that occur in patients treated with AS1986NS

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - HCA Florida Kendall Hospital, Miami, Florida
  - Icahn School of Medicine at Mount Sinai (ISMMS), New York, New York
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Background] Kommidi H, Guo H, Nurili F, Vedvyas Y, Jin MM, McClure TD, Ehdaie B, Sayman HB, Akin O, Aras O, Ting R. 18F-Positron Emitting/Trimethine Cyanine-Fluorescent Contrast for Image-Guided Prostate Cancer Management. J Med Chem. 2018 May 10;61(9):4256-4262. doi: 10.1021/acs.jmedchem.8b00240. Epub 2018 Apr 20. PMID 29676909
- [Background] Guo H, Kommidi H, Vedvyas Y, McCloskey JE, Zhang W, Chen N, Nurili F, Wu AP, Sayman HB, Akin O, Rodriguez EA, Aras O, Jin MM, Ting R. A Fluorescent, [18F]-Positron-Emitting Agent for Imaging Prostate-Specific Membrane Antigen Allows Genetic Reporting in Adoptively Transferred, Genetically Modified Cells. ACS Chem Biol. 2019 Jul 19;14(7):1449-1459. doi: 10.1021/acschembio.9b00160. Epub 2019 Jun 17. PMID 31120734
- [Background] Aras O, Demirdag C, Kommidi H, Guo H, Pavlova I, Aygun A, Karayel E, Pehlivanoglu H, Yeyin N, Kyprianou N, Chen N, Harmsen S, Sonmezoglu K, Lundon DJ, Oklu R, Ting R, Tewari A, Akin O, Sayman HB. Small Molecule, Multimodal, [18F]-PET and Fluorescence Imaging Agent Targeting Prostate-Specific Membrane Antigen: First-in-Human Study. Clin Genitourin Cancer. 2021 Oct;19(5):405-416. doi: 10.1016/j.clgc.2021.03.011. Epub 2021 Mar 19. PMID 33879400